CLINICAL TRIAL: NCT01198314
Title: Gradual Withdrawal of Immunosuppression in Long Term Stable Liver Transplant Recipients Using Immunologic Profile Predicting Operational Tolerance
Brief Title: Withdrawal of Immunosuppression in Long Term Stable Liver Transplant Recipients
Acronym: tolerance
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: liver transplantation unit, Seoul St. Mary's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCLTIT; A092258-0911-1030100 (Other Grant/Funding Number: A092258-0911-1030100)
Record Dates: First submitted 2010-09-07; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-07

CONDITIONS: Liver Transplantation
Keywords: long term; stable; recipients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LT, withdrawal of immunosuppression (Experimental)
  Interventions: Procedure: immunosuppression withdrawal
- LT, maintenance of immunosuppression (Active Comparator)
  Interventions: Procedure: continue of taking immunosuppressant

INTERVENTIONS:
Procedure: immunosuppression withdrawal — tapering off immunosuppressant
  Other Names: WIS
  Arms: LT, withdrawal of immunosuppression
Procedure: continue of taking immunosuppressant — maintain immunosuppression
  Other Names: MIS
  Arms: LT, maintenance of immunosuppression

SUMMARY:
Long-term immunosuppression carries potential adverse effects such as risk of infection, malignancy, renal insufficiency, diabetes and hypertension. In clinical liver transplantation, some liver transplant recipients maintain allograft function without immunosuppressive drugs. This is called as "operational tolerance". Many attempts have been made to identify immunological biomarkers predicting operational tolerant patients. Therefore, the investigators aimed to identify patients who have the potential to be operationally tolerant using biomarkers, withdraw immunosuppressant gradually and stop ultimately with monitoring of biomarkers.

DETAILED DESCRIPTION:
Among long term stable liver transplant recipients, we will select some proportion of patients who have the high potential for obtaining operational tolerance using biomarkers.

Then, we will gradually reduce immunosuppressants and monitor biomarkers as well as biochemical tests. The course of tapering off immunosuppressant will take about 1 year.

During withdrawal of immunosuppression, participants will be closely monitored for liver enzyme, immunological profile.

If there are some signs of rejection, liver biopsy will be undertaken and participants will be treated using immunosuppressant.

After complete withdrawal of immunosuppressant, participants will be followed for at least of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* long term stable liver transplant recipients

Exclusion Criteria:

* liver transplant due to autoimmune disease
* liver transplant due to hepatitis C virus (HCV)
* history of graft rejection
* history of biliary infection or stricture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
number of participants who have the potential for the operational tolerance | in the 2 years fololowing study enrollment
  measure number of patients who can be weaned off immunosuppression completely

SECONDARY OUTCOMES:
Tolerance biomarker | 1 year following immunosuppression withdrawal
  find out biomarkers which can predict operational tolerance
immunologic profile related to rejection | up to 2 years following withdrawal of immunosuppression
  observe immunologic profile changes which are related to rejection

CONTACTS AND LOCATIONS:
Overall Officials: Jong Young Choi, Professor, Study Chair — The Catholic University of Korea
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

REFERENCES:
- [Background] Castellaneta A, Thomson AW, Nayyar N, de Vera M, Mazariegos GV. Monitoring the operationally tolerant liver allograft recipient. Curr Opin Organ Transplant. 2010 Feb;15(1):28-34. doi: 10.1097/MOT.0b013e328334269a. PMID 19890211